CLINICAL TRIAL: NCT02541071
Title: Influence of the Noradrenergic System on the Formation of Intrusive Memories: An Experimental Approach With a Trauma Film Paradigm
Brief Title: Influence of the Noradrenergic System on the Formation of Intrusive Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dipl.- Psych. Felicitas Rombold, Dipl.-Psych., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Rombold_01
Record Dates: First submitted 2015-08-06; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Intrusive Memories
MeSH Terms: interventions — Yohimbine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yohimbine and Stress Film (Experimental): Administration of 10mg yohimbine before the trauma film.
  Interventions: Behavioral: Stress Film; Drug: Yohimbine
- Placebo and Stress Film (Experimental): Administration of placebo before the trauma film.
  Interventions: Behavioral: Stress Film; Drug: placebo
- Clonidine and Stress Film (Experimental): Administration of 0.15mg clonidine before the trauma film.
  Interventions: Behavioral: Stress Film; Drug: Clonidine

INTERVENTIONS:
Behavioral: Stress Film
Drug: Yohimbine
  Arms: Yohimbine and Stress Film
Drug: Clonidine
  Arms: Clonidine and Stress Film
Drug: placebo
  Arms: Placebo and Stress Film

SUMMARY:
Intrusive memories of traumatic events are core features of posttraumatic stress disorder (PTSD) but little is known about the neurobiological formation of intrusions. The aim of this study was to determine whether the activity of the noradrenergic system during an intrusion-inducing stressor influences subsequent intrusive memories.

DETAILED DESCRIPTION:
The investigators conducted an experimental, double-blind, placebo-controlled study in 118 healthy women. Prior to watching an established trauma film paradigm that induces short lasting intrusions, participants received a single dose of either 10 mg yohimbine, stimulating noradrenergic activity, or 0.15 mg clonidine, inhibiting noradrenergic activity, or placebo. The number of consecutive intrusions of the trauma film, the mean vividness of the intrusions and the mean degree of distress evoked by the intrusions were assessed during the following four days. Salivary cortisol and alpha-amylase were collected at seven time points prior to, and after the trauma film.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* German on a native level

Exclusion Criteria:

* former or present DSM IV Axis I disorders
* physical illnesses
* any medication intake (except oral contraceptive)
* history of sexual abuse or rape
* pregnancy or lactation period

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories | four consecutive days
  Measured with an intrusion diary

SECONDARY OUTCOMES:
Vividness of intrusive memories | four consecutive days
  Measured with an intrusion diary
Degree of distress of intrusive memories | four consecutive days
  Measured with an intrusion diary

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, Dr., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité University Medicine Berlin, Campus Benjamin Franklin, Berlin, State of Berlin, Germany